CLINICAL TRIAL: NCT00171145
Title: A 12-Week Study to Evaluate the Efficacy of Darifenacin to Increase the Warning Time in Patients With Overactive Bladder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDAR328A2401
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder, incontinence, antimuscarinic, warning time, darifenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin — Darifenacin 15 mg tablets once daily
  Other Names: Enablex
  Arms: 1
Drug: Placebo — Placebo tablets once daily
  Arms: 2

SUMMARY:
This study will assess the efficacy of a 12-week treatment with darifenacin in increasing warning time, the time from first sensation of urgency to voiding, in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Three symptoms of OAB (urge incontinence, frequency and urgency) for at least six months prior to Visit 2.
* Patients capable of independent toileting and able of independently completing the patient diary.

Exclusion Criteria:

* Patients in whom the use of anticholinergic drugs was contraindicated
* Evidence of severe liver disease
* Patients with other clinically significant urinary or gynecological conditions

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2004-04; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in warning time at week 12.

SECONDARY OUTCOMES:
Change in warning time at weeks 2 & 6.
Change in frequency of urge incontinence episodes.
Change in frequency of micturitions.
Change in mean volume per void.
Change in frequency of urgency.
Safety and tolerability.
Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Novartis, East Hanover, New Jersey, United States